CLINICAL TRIAL: NCT01748357
Title: Pattern Recognition of Volatile Organic Compounds (VOC) in Exhaled Breath for the Diagnosis of Pulmonary Tuberculosis
Brief Title: Siemens VOC TB Pilot Study
Status: Completed | Type: Observational
Sponsor: Research Center Borstel (Other)
Collaborators: Siemens Corporate Technologies (Unknown)
Responsible Party: Principal Investigator, Christian Herzmann, Head of Center for Clinical Trials, Research Center Borstel
Other Study IDs: RCBorstel003
Record Dates: First submitted 2012-12-07; First posted 2012-12-12 (Estimated); Last update posted 2014-11-06 (Estimated); Status verified 2014-11

CONDITIONS: Tuberculosis
Keywords: Tuberculosis; Volatile organic compounds; exhaled breath; Siemens
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Volatile compounds from exhaled breath
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Tuberculosis group: Patients with confirmed pulmonary infection with M. tuberculosis. At least 50% of the subjects should be tested before therapy is started. Patients with treatment for tuberculosis >1 week are excluded.
- Inflammation group: Patients with another inflammatory disease of the lower respiratory tract, i.e. pneumonia, sarcoid or bronchial carcinoma. This group is required to detect VOC pattern caused by pulmonary inflammation.
- Healthy group: Healthy subjects without lung disease. These subjects should be recruited from outside the hospital / study site to avoid confounding VOC pattern caused by continuous exposure to the hospital environment.

SUMMARY:
Tuberculosis is a bacterial infection causing 1.1 million deaths annually worldwide. Diagnosis of the disease is often time consuming or challenging. Many cases of tuberculosis require advanced and expensive diagnostic methods that restrict their availability in resource limited countries where the burden of tuberculosis is highest. The development of rapid point of care diagnostics is required.

Published data confirm that trained African giant-pouched rats are able to identify M. tuberculosis cultures through olfactory recognition. A first trial using an electronic nose reported a rate of detection of 85% in tuberculosis patients. A further trial was closed in June 2011 but remains unpublished, yet. The olfactory pattern that potentially allows the recognition of tuberculosis remains unknown.

This trial aims to detect first patterns of volatile organic compounds (VOCs) that bear a potential for further development and fine tuning. A technical prototypic device of Siemens is used for pattern detection.

The study is comparing 3 groups of patients:

* patients with confirmed active pulmonary tuberculosis (n=20)
* patients with other inflammatory lung diseases (pneumonia, sarcoidosis, COPD, bronchial carcinoma) (n=20)
* healthy volunteers that do not work in the hospital or visit the hospital regularly Detailed data for all study subjects will be collected for this trial in order to eliminate confounding factors. Furthermore, detailed data of the surroundings of the patient, the surroundings of the technical device and of the operator will be captured.

Hypothesis:

The pattern of exhaled volatile organic compounds allows the detection of pulmonary tuberculosis

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed pulmonary infection with M. tuberculosis (MTB) or other inflammatory disease of the lower respiratory tract (i.e. pneumonia, sarcoid, bronchial carcinoma) or healthy subject that is not employed or working at the study site
2. Oral and written consent to study participation

Exclusion Criteria:

1. Tuberculosis therapy >1 week
2. Inability to follow the study requirements
3. Patient in custodianship or guardianship
4. Other lung diseases that are not listed in the inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: See groups described above
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2012-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Percentage of correctly identified patients with tuberculosis | Day of admission to hospital
  The VOC pattern is used to differentiate tuberculosis patients from patients with non-tuberculosis inflammatory lung disease and from healthy volunteers

SECONDARY OUTCOMES:
Change in VOC pattern induced by storage for several days | At days 3, 5 and 7 after sample collection
Change in VOC pattern induced by storage temperature | At days 3, 5 and 7 after sample collection
Change in VOC pattern induced by tuberculosis therapy | After completion of recruitment

CONTACTS AND LOCATIONS:
Locations (1):
- Research Center Borstel, Borstel, Schleswig-Holstein, Germany